CLINICAL TRIAL: NCT00184574
Title: Comparison of the Effect on Glycemic Control of Biphasic Insulin Aspart 70/30, Biphasic Insulin Aspart 50/50, and Biphasic Insulin Aspart 30/70 All in Combination With Metformin in Subjects With Type 2 Diabetes (the INTENSIMIX Trial).
Brief Title: Comparison of Biphasic Insulin Aspart 70/30, 50/50, and 30/70 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1440
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: metformin

SUMMARY:
This trial is conducted in Europe. This trial aims for a comparison of the effect on glycemic control in subjects with type 2 diabetes of three different premixed insulin analogues given in combination with an oral anti-diabetic drug.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with insulin
* Currently treated with Metformin
* HbA1c: 7.5-12.0%

Exclusion Criteria:

* Body Mass Index (BMI) < 25.0 or > 40.0 kg/m2
* Metformin contraindications according to local practice
* TZDs within 6 months prior to randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2005-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 36 weeks

SECONDARY OUTCOMES:
8-point plasma glucose profiles
Safety variables
Other glycemic variables

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (103):
- Austria (5):
  - Novo Nordisk Investigational Site, Bregenz
  - Novo Nordisk Investigational Site, Feldkirch
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Belgium (5):
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Genk
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Liège
- Bulgaria (2):
  - Novo Nordisk Investigational Site, Pleven
  - Novo Nordisk Investigational Site, Sofia
- Czechia (3):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Prague
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Køge
  - Novo Nordisk Investigational Site, Odense
- France (11):
  - Novo Nordisk Investigational Site, Antibes
  - Novo Nordisk Investigational Site, Boulogne-Billancourt
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Chesnay
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Metz
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Perpignan
- Germany (15):
  - Novo Nordisk Investigational Site, Bad Heilbrunn
  - Novo Nordisk Investigational Site, Beckum
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Genthin
  - Novo Nordisk Investigational Site, Kippenheim
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Saarbrücken
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Schönebeck
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Würzburg
- Hungary (3):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Veszprém
- Italy (11):
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Gazi
  - Novo Nordisk Investigational Site, Lucca
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Salerno
  - Novo Nordisk Investigational Site, Savigliano (CN)
  - Novo Nordisk Investigational Site, Terni
  - Novo Nordisk Investigational Site, Udine
- Netherlands (6):
  - Novo Nordisk Investigational Site, 's-Hertogenbosch
  - Novo Nordisk Investigational Site, Amersfoort
  - Novo Nordisk Investigational Site, Brunssum
  - Novo Nordisk Investigational Site, Hoogeveen
  - Novo Nordisk Investigational Site, Roosendaal
  - Novo Nordisk Investigational Site, Rotterdam
- Poland (6):
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Mazowieckie
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Romania (4):
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Galati
  - Novo Nordisk Investigational Site, Suceava
  - Novo Nordisk Investigational Site, Târgu Mureş
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- Spain (9):
  - Novo Nordisk Investigational Site, Albacete
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, L'Hospitalet de Llobregat
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Mostoles - Madrid -
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, San Juan
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Zaragoza
- Switzerland (5):
  - Novo Nordisk Investigational Site, Biel
  - Novo Nordisk Investigational Site, Interlaken-Unterseen
  - Novo Nordisk Investigational Site, Sankt Gallen
  - Novo Nordisk Investigational Site, Winterthur
  - Novo Nordisk Investigational Site, Zurich
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Bursa
  - Novo Nordisk Investigational Site, Istanbul
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Brighton
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cosham
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Watford

REFERENCES:
- [Result] Garber AJ, Ligthelm R, Christiansen JS, Liebl A. Premixed insulin treatment for type 2 diabetes: analogue or human? Diabetes Obes Metab. 2007 Sep;9(5):630-9. doi: 10.1111/j.1463-1326.2006.00654.x. PMID 17697056
- [Result] Cucinotta D, Smirnova O, Christiansen JS, Kanc K, le Devehat C, Wojciechowska M, Lopez de la Torre M, Liebl A. Three different premixed combinations of biphasic insulin aspart - comparison of the efficacy and safety in a randomized controlled clinical trial in subjects with type 2 diabetes. Diabetes Obes Metab. 2009 Jul;11(7):700-8. doi: 10.1111/j.1463-1326.2009.01035.x. Epub 2009 May 19. PMID 19476479
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com